CLINICAL TRIAL: NCT05546320
Title: COMParison of the EffecT of mEdication Therapy: Anticoagulation Versus Anti-platelet Versus Migraine Therapy in Alleviating Migraine With Patent Foramen Ovale
Brief Title: Comparison of the Effect of Medication Therapy in Alleviating Migraine With Patent Foramen Ovale
Acronym: COMPETE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Project Manager, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No2022-1758
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Patent Foramen Ovale; Migraine
Keywords: Migraine; Patent Foramen Ovale; Medication therapy
MeSH Terms: conditions — Foramen Ovale, Patent; Migraine Disorders | interventions — Aspirin; Metoprolol; Tablets; Clopidogrel; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Migraine Medication Group (Active Comparator): Patients randomized into migraine medication group will be given Metoprolol 25mg twice a day as the control group.
  Interventions: Drug: Metoprolol 25 Mg Oral Tablet
- Anticoagulation or anti-platelet medication Group 1 (Experimental): Patients randomized into anticoagulation or anti-platelet medication group will be given aspirin.
  Interventions: Drug: Aspirin 100mg
- Anticoagulation or anti-platelet medication Group 2 (Experimental): Patients randomized into anticoagulation or anti-platelet medication group will be given clopidogrel.
  Interventions: Drug: Clopidogrel 75mg
- Anticoagulation or anti-platelet medication Group 3 (Experimental): Patients randomized into anticoagulation or anti-platelet medication group will be given Rivaroxaban.
  Interventions: Drug: Rivaroxaban 20mg

INTERVENTIONS:
Drug: Aspirin 100mg — Anticoagulation or anti-platelet or migraine medication therapy will be provided for different groups.
  Arms: Anticoagulation or anti-platelet medication Group 1
Drug: Metoprolol 25 Mg Oral Tablet — Metoprolol 25mg will be provided for the participants twice a day.
  Arms: Migraine Medication Group
Drug: Clopidogrel 75mg — Clopidogrel 75mg will be provided for the participant once a day.
  Arms: Anticoagulation or anti-platelet medication Group 2
Drug: Rivaroxaban 20mg — Rivaroxaban 20mg will be provided for the participant once a day.
  Arms: Anticoagulation or anti-platelet medication Group 3

SUMMARY:
Migraine attack is an episodic disorder that affects approximately 12% of the population. Previous studies have shown that 41-48% of migraineur have a combination of patent foramen ovale (PFO). Clinical observational studies have been linking medication therapies which include anticoagulation and anti-platelet therapy with the effectiveness in improving migraine symptoms and reducing the frequency of attacks in patients combined with a PFO. However, it has been unclear whether the effectiveness of anticoagulation or anti-platelet therapy outweigh the conventional migraine medication therapy, as a result, we designed a multi-center randomized clinical trial aiming to examine the effectiveness of anticoagulation versus anti-platelet versus migraine medication therapy in migraine patients with PFO and provide a clinical guidance for migraineur.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 ；
2. Diagnosed migraine by ICHD-3
3. History of migraine longer than 1 year
4. TCD/TTE/TEE diagnosed patent foramen ovale
5. Willing to participant and agree to follow-ups

Exclusion Criteria:

1. Migraine caused by other reason
2. Had TIA/stroke history
3. Hypersensitive or hyposensitive to the study drug
4. With a history of anticoagulation or anti-platelet drug intake 3 month before randomization.
5. With a history of metoprolol intake 3 month before randomization, and migraine attacks did not reduced 50%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Responder rate | From baseline period to 3-month treatment period
  Defined as a 50% reduction from the monthly number of migraine attacks during the baseline phase to the monthly number of migraine attacks during the treatment phase.
Treatment safety | From baseline period to 3-month treatment period
  Adverse events after medication treatment

SECONDARY OUTCOMES:
Migraine days change per month | From baseline period to 3-month treatment period
  Change in the mean number of migraine days from baseline to treatment phase.
Number of migraine attacks change per month | From baseline period to 3-month treatment period
  Change in the mean number of migraine attacks from baseline to treatment phase.
Percentage of migraine change | From baseline period to 3-month treatment period
  Participants experienced 75%, or greater reduction in migraine headache attacks during treatment phase as compared to baseline phase.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Z, Dong J, Yan Y, Fang F, Wang C, Zhang F, Ouyang W, Wang S, Pan X. Study design and rationale of COMPETE: Comparison of the effect of medication therapy in alleviating migraine with patent foramen ovale. Am Heart J. 2024 Mar;269:1-7. doi: 10.1016/j.ahj.2023.12.011. Epub 2023 Dec 16. PMID 38109984